CLINICAL TRIAL: NCT00279370
Title: Antidepressant Use During Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Wisner, Professor of Psychiatry, Obstetrics and Gynecology and Reproductive Sciences, Epidemiology and Women's Studies, University of Pittsburgh
Other Study IDs: R01MH060335 (NIH); R01MH060335 (NIH); DSIR AT-SO
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Depression
Keywords: SSRI Exposure; Pregnancy; Infant Development
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will determine the safety of antidepressant use during pregnancy for both the mother and the child.

DETAILED DESCRIPTION:
Symptoms of major depressive disorder (MDD) include persistent sad mood, feelings of hopelessness or guilt, decreased energy, irritability, and more. If untreated, MDD can interfere with the ability to work, study, sleep, eat, and enjoy once pleasurable activities. MDD occurs most commonly in females between the ages of 25 and 44. This puts women of childbearing age at a particularly high risk for developing the disorder. However, very little research has been done to determine the safety of antidepressant use during pregnancy and how the medication may affect the baby. This study will determine the safety of antidepressant use during pregnancy for both the mother and the child.

Participants in this observational study will not receive medication or treatment of any kind. Pregnant woman who are already taking medication for depression will be recruited, in addition to pregnant women who are not taking any medication. The participants will first undergo interviews to establish their psychiatric diagnoses. Subsequent interviews will be held to monitor levels of depressive symptoms, exposure to other substances that could potentially harm the fetus, levels of antidepressants in the blood, and dietary intake during pregnancy. Participants will report to the study site for these evaluations at Weeks 20, 30, and 36 of pregnancy. From Week 36 to Week 40, interviews will be conducted over the phone.

At birth, cord blood will be collected and the infant's cries will be recorded. The infant's development will be assessed at 2 weeks and 3, 6 ½, 12, 18, and 24 months postpartum. Mothers who take selective serotonin reuptake inhibitors (SSRIs) and are breastfeeding their children will report to the study site with their children at 1 month postpartum to measure the level of SSRIs in the infant's blood. In addition, digital photographs of the infant's face, profile, hands, and torso will be taken at 2 weeks and 3, 12, and 24 months postpartum. Additional face-only photographs of the infant will be taken at these times and at birth for further in-depth analyses of facial characteristics. Mother-child interactions will be videotaped at all postpartum assessments.

ELIGIBILITY:
Inclusion Criteria:

* Less than 24 weeks pregnant at the time of study entry
* As of 12/1/2005, at significant risk for developing depression or currently taking SSRIs during pregnancy

Exclusion Criteria:

* History of or current psychosis, bipolar disorder, or schizoaffective disorder
* Current substance use disorder
* Any medical condition that may be related to outcomes (such as multiple births or insulin-dependent diabetes)
* Has not attended at least two prenatal visits at the 20-week intake point

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with or without active depression and with or without SSRI use in pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 1999-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
SIGH-ADS | 20, 30, 36 weeks gestation and 2, 12, 28, 52, and 104 weeks postpartum
Bayley Scales of Infant Development | 12, 28, 52, and 104 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L. Wisner, MD MS, Principal Investigator — University of Pittsburgh, Department of Psychiatry
Locations (1):
- Women's Behavioral HealthCARE Program, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Gollan JK, Yang A, Ciolino JD, Sit D, Wisner KL. Postpartum anhedonia: Emergent patterns in bipolar and unipolar depression. Psychiatry Res. 2021 Dec;306:114274. doi: 10.1016/j.psychres.2021.114274. Epub 2021 Nov 9. PMID 34837882
- [Derived] Wisner KL, Sit D, O'Shea K, Bogen DL, Clark CT, Pinheiro E, Yang A, Ciolino JD. Bipolar disorder and psychotropic medication: Impact on pregnancy and neonatal outcomes. J Affect Disord. 2019 Jan 15;243:220-225. doi: 10.1016/j.jad.2018.09.045. Epub 2018 Sep 18. PMID 30248632
- [Derived] Yang A, Ciolino JD, Pinheiro E, Rasmussen-Torvik LJ, Sit DKY, Wisner KL. Neonatal Discontinuation Syndrome in Serotonergic Antidepressant-Exposed Neonates. J Clin Psychiatry. 2017 May;78(5):605-611. doi: 10.4088/JCP.16m11044. PMID 28570796
- [Derived] Kim DR, Pinheiro E, Luther JF, Eng HF, Dills JL, Wisniewski SR, Wisner KL. Is third trimester serotonin reuptake inhibitor use associated with postpartum hemorrhage? J Psychiatr Res. 2016 Feb;73:79-85. doi: 10.1016/j.jpsychires.2015.11.005. Epub 2015 Nov 19. PMID 26692255
- [Derived] Santucci AK, Singer LT, Wisniewski SR, Luther JF, Eng HF, Dills JL, Sit DK, Hanusa BH, Wisner KL. Impact of prenatal exposure to serotonin reuptake inhibitors or maternal major depressive disorder on infant developmental outcomes. J Clin Psychiatry. 2014 Oct;75(10):1088-95. doi: 10.4088/JCP.13m08902. PMID 25373117
- [Derived] Sit D, Perel JM, Wisniewski SR, Helsel JC, Luther JF, Wisner KL. Mother-infant antidepressant concentrations, maternal depression, and perinatal events. J Clin Psychiatry. 2011 Jul;72(7):994-1001. doi: 10.4088/JCP.10m06461. PMID 21824458
- [Derived] Sit D, Perel JM, Luther JF, Wisniewski SR, Helsel JC, Wisner KL. Disposition of chiral and racemic fluoxetine and norfluoxetine across childbearing. J Clin Psychopharmacol. 2010 Aug;30(4):381-6. doi: 10.1097/JCP.0b013e3181e7be23. PMID 20631556
- [Derived] Wisner KL, Sit DK, Hanusa BH, Moses-Kolko EL, Bogen DL, Hunker DF, Perel JM, Jones-Ivy S, Bodnar LM, Singer LT. Major depression and antidepressant treatment: impact on pregnancy and neonatal outcomes. Am J Psychiatry. 2009 May;166(5):557-66. doi: 10.1176/appi.ajp.2008.08081170. Epub 2009 Mar 16. PMID 19289451
- [Derived] Sit DK, Perel JM, Helsel JC, Wisner KL. Changes in antidepressant metabolism and dosing across pregnancy and early postpartum. J Clin Psychiatry. 2008 Apr;69(4):652-8. doi: 10.4088/jcp.v69n0419. PMID 18426260